CLINICAL TRIAL: NCT03009747
Title: A Prospective, Randomization and Clinic Cohort Observational Study From Multi Institutions on Bowel Dysfunction Following Surgery for Rectal Cancers With Sphincter Preservation
Brief Title: A Prospective Multi-Center Research on Bowel Dysfunction After Sphincter Preservative Surgery
Acronym: PMCRBDSPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First People's Hospital of Changzhou (Other); Peking University Cancer Hospital & Institute (Other); Beijing Friendship Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Hebei Medical University Fourth Hospital (Other); First Affiliated Hospital of Jiamusi University (Unknown); China-Japan Friendship Hospital (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other); Xiangya Hospital of Central South University (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Peking University International Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BaS-1611
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Bowel Dysfunction; Rectal Cancer
Keywords: rectal cancer; anterior resection syndrome; sphincter-preserving surgery
MeSH Terms: conditions — Intestinal Diseases; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sphincter-preserving surgery: Patients meet the inclusion criteria will be enrolled into this observing group

SUMMARY:
This research plans to collect rectal cancer patients after sphincter-preserving surgery from 14 institutions in China mainland, observe the incidence and risk factors about bowel dysfunction after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Adenocarcinoma confirmed by pathology
3. Distance from the lowest margin of tumor to the anal verge is ≤ 12cm, confirmed by hard sigmoidoscope.
4. The tumor is estimated to be resectable and confirmed by multidisciplinary team (MDT).
5. The operation is estimated to be sphincter-preserving.
6. The Eastern Cooperative Oncology Group(ECOG) performance status score of patient is ≤ 2.
7. The estimated life time is not less than one year.
8. The patient agree to sign the informed consent.

Exclusion Criteria:

1. The patient refuse to follow research plan.
2. Emergency case
3. Pregnant and lactating female patient
4. The patient did not accept radical resection.
5. The patient did not accept first stage resection and anastomosis.
6. The patient has experienced anal-rectal surgery.
7. The patient has experienced left colon surgery.
8. The patient suffered long-existing bowel dysfunction before rectal cancer diagnosis.
9. The patient was diagnosed with cognitive or communicative obstacles.
10. The patient was diagnosed with serious repeated infection or other concomitance diseases.
11. The patient has participated other medical research which may affect his/her bowel function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients who accept sphincter-preserving surgery
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of bowel dysfunction after sphincter-preserving surgery | one year
Risk factors of bowel dysfunction after sphincter-preserving surgery | one year

SECONDARY OUTCOMES:
Incidence of each symptoms of bowel dysfunction | one year
Prognosis of bowel dysfunction after sphincter-preserving surgery | one year
Incidence of bowel dysfunction after sphincter-preserving surgery | one year
  comparing incidences between high and low anastomsis site

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, M.D./ PhD, Study Chair — Chinese Society of Colon and Rectal Surgeons

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu F, Guo P, Su X, Cui M, Jiang J, Wang S, Yu Z, Zhou R, Ye Y. A Novel Remote Follow-Up Tool Based on an Instant Messaging/Social Media App for the Management of Patients With Low Anterior Resection Syndrome: Pilot Prospective Self-Control Study. JMIR Mhealth Uhealth. 2021 Mar 19;9(3):e22647. doi: 10.2196/22647. PMID 33739295